CLINICAL TRIAL: NCT04519112
Title: Department of Cardiology, Shanghai Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Brief Title: Remote Magnetic Versus Manual Navigation-guided Ablation for Non-outflow Tract Premature Ventricular Contractions: a Prospective, Randomized, Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200001
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Premature Ventricular Contraction
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote magnetic navigation group (Experimental): PVC ablation with RMN
  Interventions: Procedure: Catheter Ablation
- Mannual control navigation group (Active Comparator): PVC ablation with mannual navigation
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Catheter Ablation — Catheter Ablation with RMN and MCN

SUMMARY:
This prospective, randomized, controlled trial is designed to compare the safety and efficacy of remote magnetic navigation-guided ablation for ventricular premature complexes arising from non-outflow tracts with manual control navigation.

ELIGIBILITY:
Inclusion Criteria:

1. non-outflow tract PVCs
2. Holter>10,000/24h or PVCs load>10%
3. the first ablation procedure
4. failure of at least one AAD to treat PVCs before ablation

Exclusion Criteria:

1. PVC ablation history
2. HF with NYHA IV
3. 3 months prior to AMI or PCI
4. Cardiac thrombosi
5. Hyperthyroidism
6. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Freedom rate of PVC | one year
  Efficacy endpoint
Procedure-related Complications | one year
  Safety endpoint

SECONDARY OUTCOMES:
fluoroscopic time | one day
ablation time | one day
procedure time | one day

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Noten AME, Hendriks AA, Yap SC, Mol D, Bhagwandien R, Wijchers S, Kardys I, Khan M, Szili-Torok T. Contact feedback improves 1-year outcomes of remote magnetic navigation-guided ischemic ventricular tachycardia ablation. Int J Cardiol. 2020 Sep 15;315:36-44. doi: 10.1016/j.ijcard.2020.05.028. Epub 2020 May 12. PMID 32413467
- [Result] Qiu X, Zhang N, Luo Q, Liu A, Ji Y, Ye J, Lin C, Ling T, Chen K, Pan W, Zhao J, Jin Q, Wu L. Remote magnetic navigation facilitates the ablations of frequent ventricular premature complexes originating from the outflow tract and the valve annulus as compared to manual control navigation. Int J Cardiol. 2018 Sep 15;267:94-99. doi: 10.1016/j.ijcard.2018.03.105. PMID 29957265